CLINICAL TRIAL: NCT06428201
Title: The Efficacy of Tele Rehabilitation- Based Task-Specific Training for Cognitive Function Improvement in Multiple Sclerosis (MS) Patients
Brief Title: The Efficacy of Tele Rehabilitation- Based Task-Specific Training for Cognitive Function Improvement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/711
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Sclerosis, Multiple
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Control Group
- EXP group (Experimental)
  Interventions: Combination Product: Experimental Group

INTERVENTIONS:
Diagnostic Test: Control Group — The control group receives standard care, which includes routine medical management and general physical rehabilitation exercises. This involves regular consultations with healthcare providers and exercises aimed at maintaining mobility and physical function. The control group also follows a schedule of three 45-minute sessions per week for 12 weeks, ensuring a consistent comparison with the experimental group.
  Arms: Control Group
Combination Product: Experimental Group — The experimental intervention involves tele-rehabilitation-based task-specific training to enhance cognitive functions in multiple sclerosis (MS) patients. This program includes cognitive exercises targeting memory, attention, executive function, and processing speed, conducted remotely via a tele-rehabilitation platform. Patients participate in three 45-minute sessions per week for 12 weeks. Each session is guided by a trained therapist, ensuring personalized support and real-time feedback.
  Arms: EXP group

SUMMARY:
"This study investigates the feasibility of tele-rehabilitation combined with targeted training for cognitive enhancement in individuals with Multiple Sclerosis (MS). Multiple sclerosis (MS) is a chronic illness that affects the central nervous system, often resulting in cognitive impairments that significantly impact quality of life. Tele-restoration provides an accessible and effective method for delivering therapeutic interventions, particularly beneficial for those with mobility limitations.

DETAILED DESCRIPTION:
The study was a randomized controlled trial with multiple sclerosis patients divided into two groups: one receiving tele-rehabilitation-based task-specific training and the other receiving conventional care. The mediation group participated in structured cognitive training sessions conducted using a tele-rehabilitation platform, focusing on tasks designed to enhance memory, attention, and executive functions. Psychological assessments were conducted during the mediation period to measure improvements.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of MS confirmed by a neurologist.
* Between 18 and 65 years of age.
* Presence of psychosis confirmed by standardized psychometric testing.
* A stable treatment environment that allows intervention.
* Internet access with camera and computer/tablet.
* Ability to understand and follow course directions.
* Willingness to give informed consent.

Exclusion Criteria:

* Severe psychiatric co-morbidities affecting cognitive function.
* Concurrent intervention with other psychological rehabilitation programs.
* Lack of availability or use of technology necessary for tele-rehabilitation.
* Further research interventions.
* Unstable medical condition

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) scale | 12 Months
  The MoCA scale is a comprehensive tool designed to evaluate various cognitive domains, including attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation. It provides a detailed assessment of cognitive performance, making it an ideal measure for tracking cognitive improvements in MS patients participating in the tele-rehabilitation and task-specific training programs.

CONTACTS AND LOCATIONS:
Locations (1):
- District Head Quarters Hospital Narowal, Circular Road, Near Jassar Bypass, Narowal Location: Khalid Eye & Medical Care Block C Commercial Area, Jubilee Town, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No